CLINICAL TRIAL: NCT06266481
Title: Topical Dexamethasone Versus Topical Lidocaine Spray to Reduce Post-intubation Sore Throat in Shoulder Arthroscopic Surgeries: A Comparative Study
Brief Title: Topical Dexamethasone Versus Topical Lidocaine Spray to Reduce POST in Shoulder Arthroscopic Surgeries: A Comparative Study
Acronym: post
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Pharos University in Alexandria (Other)
Responsible Party: Principal Investigator, mona elsaid, lecture, Pharos University in Alexandria
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: pua04202312313157
Record Dates: First submitted 2024-01-16; First posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Postoperative Sore Throat
Keywords: Sore-throat postoperative; dexamesthsone; 10% lidocaine
MeSH Terms: interventions — Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- dexamethasone group (Active Comparator): An endotracheal tube was soaked in 8mg of dexamethasone for group I intubation
  Interventions: Drug: Topical dexamethasone
- lidocaine group (Active Comparator): 10% lidocaine was sprayed over the tube
  Interventions: Drug: 10% lidocaine was sprayed over the tube for the second group

INTERVENTIONS:
Drug: Topical dexamethasone — Patients were interviewed at 1 and 6 h after extubating for post-operative sore throat (POST). POST was assessed by a modified 4-point scale (0= no sore throat, 1= mild sore throat: complains of sore throat only on asking, 2 = moderate sore throat: complains of sore throat spontaneously, and 3 = severe sore throat: change of voice or hoarseness.
  Arms: dexamethasone group
Drug: 10% lidocaine was sprayed over the tube for the second group — Patients were interviewed at 1 and 6 h after extubating for post-operative sore throat (POST). POST was assessed by a modified 4-point scale (0= no sore throat, 1= mild sore throat: complains of sore throat only on asking, 2 = moderate sore throat: complains of sore throat spontaneously, and 3 = severe sore throat: change of voice or hoarseness.
  Arms: lidocaine group

SUMMARY:
postoperative sore throat is the most frequent side effects after anaesthesia intubation. Dexamethasone and 10% lidocaine spray used prior to surgery has shown useful in managing these complications at the moment. In order to examine the prophylactic impact of local Dexamethasone and lidocaine on postoperative sore throat, this study was conducted.

DETAILED DESCRIPTION:
postoperative sore throat is the most frequent side effects after anaesthesia intubation. Dexamethasone and 10% lidocaine spray used prior to surgery has shown useful in managing these complications at the moment. In order to examine the prophylactic impact of local Dexamethasone and lidocaine on postoperative sore throat, this study was conducted.In this study, 100 patients were intubated to undergo general anaesthesia for shoulder arthroscopy and randomised into one of two groups. An endotracheal tube was soaked in 8mg of dexamethasone for the first group intubation, while 10% lidocaine was sprayed over the tube for the second group. Following extubation, the two groups examined the severity of sore throats

ELIGIBILITY:
Inclusion Criteria:

* •Patients belonging to ASA physical status I, II

  * Patients between age18 to 50 years
  * Patients belonging to both genders.
  * patients undergoing shoulder arthroscopic surgeries.
  * Patients with fasting blood glucose <100 mg/dl or random blood sugar <140 mg/dl.

Exclusion Criteria:

* Patients who are not willing to give consent for participation in the study

  * Patients with anticipated difficult airway
  * Patients who are allergic to steroids.
  * Patients with ASA physical status III, IV
  * Diabetic patients.
  * Patients on steroids
  * Patients requiring nasogastric tube or throat pack.
  * Patients posted for head and neck surgeries.
  * patient with GERD
  * Pregnant patients
  * preexisting upper respiratory tract infection.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-05-30 (Estimated)

PRIMARY OUTCOMES:
Topical dexamethasone versus topical lidocaine spray to reduce post-intubation sore throat in shoulder arthroscopic surgeries: A comparative study | 3MONTH
  This study aimed to compare the effectiveness of topical applications of dexamethasone versus lidocaine spray in prevention sore throat.Patients will be assessed at 1 and 6 h after extubation for post-operative sore throat (POST). POST will be assessed by a modified 4-point scale (0= no sore throat, 1= mild sore throat: complains of sore throat only on asking, 2 = moderate sore throat: complains of sore throat spontaneously, and 3 = severe sore throat: change of voice or hoarseness.

CONTACTS AND LOCATIONS:
Locations (1):
- Pharos University, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lee JH, Kim SB, Lee W, Ki S, Kim MH, Cho K, Lim SH, Lee KM, Choi DN, Oh M. Effects of topical dexamethasone in postoperative sore throat. Korean J Anesthesiol. 2017 Feb;70(1):58-63. doi: 10.4097/kjae.2017.70.1.58. Epub 2016 Nov 25. PMID 28184268
- [Result] Banihashem N, Alijanpour E, Hasannasab B, Zarei A. Prophylactic Effects of Lidocaine or Beclomethasone Spray on Post-Operative Sore Throat and Cough after Orotracheal Intubation. Iran J Otorhinolaryngol. 2015 May;27(80):179-84. PMID 26082898
- [Result] Jabbar ML, Mahboba JH, Meazher N. Comparing the effectiveness of topical dexamethasone emollient, lidocaine gel, and glycerin emollient on the endotracheal tube for postoperative hoarseness of voice, sore throat, and laryngospasm. J Med Life. 2023 Jun;16(6):904-907. doi: 10.25122/jml-2022-0137. PMID 37675167